CLINICAL TRIAL: NCT03946527
Title: Exploratory Phase II Study of LAnreotide in Metastatic Pheochromocytoma/PARAganglioma (LAMPARA)
Brief Title: LAnreotide in Metastatic Pheochromocytoma / PARAganglioma (LAMPARA)
Acronym: LAMPARA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Antonio Fojo (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor-Investigator, Antonio Fojo, Professor of Medicine at the Columbia University Medical Center, Dept of Med Hematology & Onc, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS2820
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Paraganglioma; Pheochromocytoma
Keywords: advanced paraganglioma; advanced pheochromocytoma; metastatic paraganglioma; metastatic pheochromocytoma; lanreotide
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- lanreotide arm (Experimental): Patients with a histopathologically confirmed diagnosis of malignant paraganglioma or pheochromocytoma and either evidence of metastases or unresectability who meet the inclusion/exclusion criteria. Approximately 40 patients will be enrolled.
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide — Participants will receive lanreotide 120 mg deep subcutaneous injection every 4 weeks (±7 days) for 52 weeks, followed by an extension phase in which all patients will continue to receive lanreotide 120 mg injection every 4 weeks (±7 days) if there is no evidence of disease progression.
  Other Names: Somatuline Depot

SUMMARY:
The objectives of this study are:

* To assess the efficacy of lanreotide given every 4 weeks in participants with advanced or metastatic paraganglioma/ pheochromocytoma.
* To assess the toxicity and safety of lanreotide in participants with advanced or metastatic paraganglioma/ pheochromocytoma.
* To document the effects of lanreotide on markers of biochemical activity in participants with advanced or metastatic paraganglioma/ pheochromocytoma.

Primary endpoints:

• Assess efficacy by estimating the tumor growth rate while a patient is enrolled on study and comparing the growth rates on lanreotide to the pre-enrolment growth rate.

Secondary endpoints include measurement of:

* Overall survival (OS)
* Progression-free survival (PFS)
* Overall response rate (ORR) according to RECIST defined as partial response (PR) + complete response (CR)
* Magnitude of reduction in levels of 24-hour urinary metanephrines, catecholamines and magnitude of reduction in serum chromogranin A, evaluated every two months while enrolled on study.

DETAILED DESCRIPTION:
Lanreotide is FDA approved for certain kinds of neuroendocrine tumors. This study seeks to determine if lanreotide is beneficial for patients with paraganglioma/ pheochromocytoma.

Given the rarity of pheochromocytoma/paraganglioma that precludes the conduct of a randomized clinical trial in a timely manner, a novel method for assessing efficacy is being proposed. Efficacy will be assessed by estimating the tumor growth rate while a patient is enrolled on study and comparing the growth rates on lanreotide to the pre-enrollment growth rates. The method of analysis that will be used has been previously described. For this assessment a minimum of three tumor measurements will be required.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients must fulfill all of the following criteria:

1. Male or female at least 18 years of age at the time of first dosing
2. Patients must give signed informed consent before any study-related activities are conducted.
3. Patients in the United States must have given written authorization for the release of protected health information in compliance with HIPAA regulations; patients in other countries must provide appropriate authorization as needed by regulatory authorities in each country.
4. Histologically or cytologically confirmed diagnosis of malignant paraganglioma or pheochromocytoma and either evidence of metastases or unresectability.
5. Evidence of recent disease progression (radiological, biochemical, symptomatic) while the patient was either not receiving any therapy or was receiving a therapy that was deemed ineffective.
6. Measurable disease defined as that which can be measured in at least one dimension with a minimum size of 10 mm by CT scan. The patient must also have at least three baseline radiographic studies obtained in the previous twelve months with at least one scan obtained within six weeks of enrollment. If a patient being considered for enrollment on trial has not had three scans performed in the twelve months prior to enrollment and if in the opinion of the investigator a delay of one month will not impact the clinical course, then enrollment on protocol and the start of the lanreotide therapy can be delayed by one month or longer to obtain the additional time point. If in the opinion of the investigator such a delay may have adverse consequences then enrollment on the protocol should not be considered as an option
7. Confirmation of positive somatostatin receptor status (SRS) by Somatostatin Receptor Scintigraphy. Either of these studies will need to have been performed in the 6 months prior to the screening visit. Only if one has not been performed within the previous 6 months will a SRS study be required. if an SRS is required, it will be performed greater than or equal to 24 hours after a previous injection of subcutaneous octreotide).
8. Patients may not have had prior octreotide, long acting release (LAR)-octreotide, lanreotide or a therapeutic radiolabeled somatostatin analog (PRRT)
9. Eastern Cooperative Oncology Group (ECOG) 0-2.
10. Life expectancy of greater than 12 weeks.
11. Patients must have prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) within 2 x the upper limit
12. Patients may have had prior radiation therapy. A minimum of 42 days must have elapsed between the end of radiotherapy and registration onto the study. Measurable disease must exist outside of the radiation field for eligibility.
13. Previous surgery: Previous major surgery is permitted provided that it was performed at least 28 days prior to patient registration.
14. Laboratory requirements [parameter limits]: Absolute granulocyte count (AGC) greater than 1.5 x 109/L; platelet count greater than100 x 109/L; serum bilirubin less than 1.5 x upper limit of normal (ULN); serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN; serum amylase less than1.5 x ULN; serum lipase less than 1.5 x ULN; serum calcium less than 3 mmol/L; serum creatinine less than 1.5 x ULN
15. If female, the patient must not be pregnant (confirmed by negative pregnancy test) and must have the following documented via verbally given history:

    * At least 1 year postmenopausal (natural cessation of menses), or
    * Surgically sterile (if by tubal ligation, surgery must have been performed more than 3 months prior to entry into the study), or
    * If of childbearing potential and sexually active, she must be using or agree to use an acceptable form of contraception (oral, injected, transdermal or implanted contraceptives, diaphragm or barrier method with spermicidal and/or intrauterine device); local methods such as condoms or sponges/vaginal tablets are only to be used as an additional form of contraception.
16. If the male patient has a partner of childbearing potential and he is sexually active, he must be using or agree to use a barrier method of contraception (condom with spermicidal preferred).
17. Be able to communicate and cooperate with the principal investigator and the staff and willing to comply with the study instructions

Exclusion Criteria:

A patient who meets any of the following criteria is ineligible for participation in the study:

1. Patient has a history of known allergy or hypersensitivity to:

   * Investigational drug or any components of its formulation
   * Lanreotide, octreotide or any other somatostatin analog
2. Treatment with any other investigational drug or with "cytotoxic chemotherapy" within 28 days prior to the start of study therapy (lanreotide) and/or at any time during the patient's participation in the study
3. Treatment with sunitinib, radiotherapy, a radiolabelled specific somatostatin receptor (SSTR) analog, and/or tumor debulking less than 14 days prior to the start of study therapy (lanreotide). Treatment with metaiodobenzylguanidine (MIBG) therapy less than 90 days prior to the start of study therapy (lanreotide).
4. History of hepatic arterial embolization or hepatic arterial chemoembolization less than 28 days prior to the start of study therapy (lanreotide). Measurable disease shall exist outside of treated lesions for eligibility.
5. History of hepatic selective internal radiation therapy (e.g. Sir-spheres) less than 90 days prior the start of study therapy (lanreotide). Measurable disease shall exist outside the liver for eligibility.
6. Uncontrolled diabetes (defined as inability to maintain fasting blood glucose levels below 200 mg/dL despite best medical therapy, within last 28 days prior to screening) and/or hypertension (defined as inability to maintain blood pressure levels below systolic 140 mm Hg and/or diastolic 90 mm Hg on at least three antihypertensive medications, within last 28 days prior to screening).
7. Renal impairment (glomerular filtration rate less than 30 ml/min/1.73m2) and/or liver impairment (serum total bilirubin greater than 1.5 x ULN, or greater than 2.5 x ULN if liver metastases)
8. Uncontrolled cardiac disease (acute myocardial infarction, unstable angina or hospitalization for decompensation of congestive heart failure within the 28 days prior to the start of study therapy (lanreotide).
9. Any malignancies except:

   * Basal cell carcinoma of the skin
   * In situ carcinoma of the cervix
   * 2 years disease-free after curative cancer treatment (completion of surgery, adjuvant chemotherapy and/or radiation, and considered no evidence of disease from non phaeochromocytomas and paragangliomas (PPGL) malignancy)
10. Any serious medical condition that could jeopardize the safety of the patient and/or the efficacy assessments of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of tumor growth | minimum of 32 weeks, up to 48 weeks
  Efficacy will be assessed by measuring the tumor growth rate while a patient is enrolled on study and comparing the growth rates on lanreotide to the pre-enrollment growth rates. Tumor growth measured by a CT or MRI scan in pre-treatment, and minimum of three scans (prior to every 3rd visit, or every 12 weeks) in post-treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | Observed for 48 weeks (start of treatment to end of treatment).
  The length of time from the start of treatment that subjects with the disease are still alive.
Overall Response Rate (ORR) | Minimum of 8 weeks, up to 48 weeks.
  ORR is defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR). Responses are based on assessments per RECIST 1.1. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have change in short axis to less than 10 mm.
  * Partial Response (PR): At least a 30% change in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival | Up to 48 weeks.
  PFS is defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 criteria and the Kaplan-Meier curve. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.
Magnitude of change in analyte levels | Minimum of 16 weeks, up to 48 weeks.
  Biochemical response of greater than 20% change in 24-hour urinary metanephrines, catecholamines and serum chromogranin A levels compared to baseline, sustained for >12-week-period. Evaluated every two months while enrolled on study, although levels may be obtained as frequently as the investigator desires.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fojo, MD, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided